CLINICAL TRIAL: NCT06442943
Title: Impact of the Digital Multi-domain Cognitive Intervention in High-risk Populations for Dementia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Yuanjiao Yan, Principal Investigator, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: K2024-04-028
Record Dates: First submitted 2024-05-29; First posted 2024-06-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cognitive Dysfunction
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants in the intervention group received the digtal multi-domain cognitive intervention. The digital multi-domain cognitive intervention system is used to carry out various intervention activities. The activities include learning about health knowledge once a week; home-based exercise three times per week, for 30 minutes each time; art therapy once a week, for 90 minutes at a time; and cognitive training, which includes memory, attention, executive function, and visuospatial training, conducted three times per week, with each session lasting 30 minutes.
  Interventions: Behavioral: Multi-domain Cognitive Intervention
- Control group (Other): Participant in the control group reveived the health education , once a week, covering the prevention and treatment of chronic diseases in the elderly, as well as healthy lifestyles for the elderly
  Interventions: Behavioral: Multi-domain Cognitive Intervention

INTERVENTIONS:
Behavioral: Multi-domain Cognitive Intervention — * Cognitive rehabilitation includes home-based exercise, three times per week, for 30 minutes each session.
    * Cognitive stimulation involves art therapy, once a week, for 90 minutes per session.
      * Cognitive training encompasses memory, attention, executive function, and visuospatial training, conducted three times per week, with each session lasting 30 minutes.
        * Health education, once a week, covering the prevention and treatment of chronic diseases in the elderly, as well as healthy lifestyles for the elderly.

SUMMARY:
Dementia is a chronic, progressive neurodegenerative disease characterized by acquired cognitive impairment as its core manifestation. The most common type of dementia is Alzheimer's Disease (AD), also known as "Senile Dementia," accounting for 60-80% of all dementia cases. Currently, there are approximately 10 million AD patients in China, with the number showing an increasing trend year by year, imposing a heavy economic and caregiving burden on families and society. Studies have shown that AD has a clinically silent period of 15 to 20 years (SCD\MCI), where the risk of developing dementia is ten times higher than that of healthy elderly individuals. Nearly 50% of MCI patients progress to dementia within 5 years, and about 14.1% of SCD patients develop dementia within the same timeframe. Early detection, diagnosis, and intervention are currently the most effective strategies for preventing and treating AD. Therefore, this study aims to verify the intervention effect of integrated cognitive intervention in high-risk populations for senile dementia (SCD, MCI) based on the cognitive rehabilitation model through randomized controlled trials, and to analyze attrition rates, participation rates, etc., which have good research and application value.

DETAILED DESCRIPTION:
Based on the cognitive rehabilitation model, this study aims to develop a digital multimodal cognitive intervention program, and conduct feasibility studies and randomized controlled trials. The intervention includes health knowledge education, exercise intervention, art intervention, and cognitive training, etc. The feasibility, effectiveness, and safety of this intervention approach will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* MCI (refer to Peterson's diagnostic criteria) or SCD (refer to the diagnostic framework proposed by Jak bondi and Jessen et al.);
* Able to communicate normally in Mandarin;
* Certain level of comprehension and judgment abilities, aware of the purpose of the survey and consents to participate.

Exclusion Criteria:

* Patients with dementia exhibiting abnormal mental behavior;
* Individuals with severe hearing or speech impairments;
* Those with serious physical illnesses who are unable to cooperate and complete the survey.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Global cognitive function | Baseline (pre-intervention), six-month follow-up (post-intervention)
  The Chinese version of Montreal Cognitive Assessment will be used to assess the global cognitive function.The scale has a total score of 30 points, encompassing eight assessment sections: visual-spatial and executive function, naming, memory, attention, language, abstraction, delayed recall, and orientation. It involves multiple cognitive domains. A higher score indicates better cognitive functioning.

SECONDARY OUTCOMES:
Memory | Baseline (pre-intervention), six-month follow-up (post-intervention)
  The Chinese version of Auditory Verbal Learning Test will be used to assess the memory. This includes immediate memory, short-term memory, long-term memory, and recognition memory. A higher score indicates better memory performance.
Verbal fluency | Baseline (pre-intervention), six-month follow-up (post-intervention)
  The Chinese version of Verbal Fluency Test will be used to assess the verbal fluency. A higher score indicates better verbal language performance.
Naming difficulty | Baseline (pre-intervention), six-month follow-up (post-intervention)
  The Chinese version of Boston Naming Test will be used to assess the naming difficulty. The total scores range from 0 to 30, a higher score indicates better language functioning.
Executive function | Baseline (pre-intervention), six-month follow-up (post-intervention)
  The Chinese version of Shape Trail Test will be used to assess the execuite function. The shorter the usage time indicates better executive functioning.
Visuospatial skills | Baseline (pre-intervention), six-month follow-up (post-intervention)
  The Chinese version of Rey-Osterrieth Complex Figure Test will be used to assess the visuospatial skills. A higher score indicates better visual-spatial structural abilities.
Health-Promoting Lifestyle | Baseline (pre-intervention), three-month follow-up(during the intervention), six-month follow-up (post-intervention)
  The Chinese version of Health-Promoting Lifestyle Profile-II will be used to assess the health lifestyle . The total score range from 40 to 160. A higher score indicates better health lifestyle.
Abilities for health practices | Baseline (pre-intervention), three-month follow-up(during the intervention), six-month follow-up (post-intervention)
  The Chinese version of self-rated abilities for health practices scale will be used to assess the ability of health practice. The total score range from 0 to 112. A higher score indicates higher self-efficacy in healthy behaviors.
Lonliness | Baseline (pre-intervention), three-month follow-up(during the intervention), six-month follow-up (post-intervention)
  The University of California at Los Angels Loneliness scale will be used to assess the loneliness. A higher score indicates more lonliness.
Social network | Baseline (pre-intervention), three-month follow-up(during the intervention), six-month follow-up (post-intervention)
  The Lubben Social Network Scale will be used to assess the social network. The lower score indicates lower risk of social isolation.
Quality of life of Alzheimer's disease | Baseline (pre-intervention), three-month follow-up(during the intervention), six-month follow-up (post-intervention)
  The Quality of life-Alzheimer's disease scale will be used the quality of life. A higher score indicates better quality of life. The highest score is 39 points.
Anxiety | Baseline (pre-intervention), three-month follow-up(during the intervention), six-month follow-up (post-intervention)
  The Self-rating Anxiety Scale will be used to assess the anxiety. The subjects will fill in the form based on their own situation in the past week.
Depression | Baseline (pre-intervention), three-month follow-up(during the intervention), six-month follow-up (post-intervention)
  The Geriatric Depression Scale will be used to assess the depression. The Cronbach coefficient of this scale is 0.93.
Self-efficacy | Baseline (pre-intervention), three-month follow-up(during the intervention), six-month follow-up (post-intervention)
  The Chinese version of Self-efficacy Scale will be used to assess the self-efficacy. The total score range from 10 to 40.
Self-esteem | Baseline (pre-intervention), three-month follow-up(during the intervention), six-month follow-up (post-intervention)
  The Self-esteem Scale will be used to assess the self-esteem. A higher score indicates higher level of Self-esteem.
Sleep quality | Baseline (pre-intervention), six-month follow-up (post-intervention)
  The Athens Insomnia Scale will be used to assess the sleep quality.The Cronbach coefficient of this scale is 0.89, highest score is 24.
Subjective cognitive function | Baseline (pre-intervention), three-month follow-up(during the intervention), six-month follow-up (post-intervention)
  The Subjective Cognitive Decline Questionnaire 9 will be used to assess the subjective cognitive function. The Cronbach coefficient of this scale is 0.88, highest score is 9.

CONTACTS AND LOCATIONS:
Overall Officials: Yuanjiao Yan, PhD, Study Director — Shengli clinical medical college of Fujian Medical university
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
Research data and research-related materials will be available in a repository or online. After completion of the study, relevant data will be provided in the form of a universal resource locator or digital object identifier.
Supporting Information: SAP, Analytic Code
Time Frame: After completion of the study, relevant data will be provided in the form of a universal resource locator or digital object identifier.
Access Criteria: Researchers whose proposed use of the data has been approved

REFERENCES:
- [Derived] Yan Y, Lin X, Lu Y, Fang Z, Fu X, Wu S, Wei B, Wang Z, Chen Y, Chen Z, Lin R, Li H. Effects of a Digital Multidomain Cognitive Intervention in Older People at High Risk of Dementia: A Randomized Clinical Trial. J Clin Psychiatry. 2026 Jan 7;87(1):25m15860. doi: 10.4088/JCP.25m15860. PMID 41499182